CLINICAL TRIAL: NCT05349448
Title: Can Dexmedetomidine With Hyalase Augment Quality and Duration of Analgesia When Added to Lumbar Epidural Steroid in Failed Back Surgery. Randomized Double Blind Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 270/3-2022
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pain, Neuropathic
Keywords: neuropathy
MeSH Terms: conditions — Neuralgia | interventions — hylase; Triamcinolone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- solo group (Active Comparator): Bupivacaine 5 mg (1 mL) + Triamcinolone 40 mg (1 mL) + Saline solution (2 mL) + Hyaluronidase 1,500 IU reconstituted in 1 mL distilled water (HYL)
  Interventions: Drug: Hylase plus Triamcinolone plus sterile isotonic saline
- dex plus hyalase group (Active Comparator): Bupivacaine 5 mg (1 mL) + Triamcinolone 40 mg (1 mL) + Dexmedetomidine 0.5mic/kg + Hyaluronidase 1,500 IU reconstituted in 1 mL distilled water (HYL)+ Saline solution (2 mL)
  Interventions: Drug: Hylase plus Dexmedetomidine plus Triamcinolone

INTERVENTIONS:
Drug: Hylase plus Triamcinolone plus sterile isotonic saline — transforaminal fluroscopic epidural injection
  Arms: solo group
Drug: Hylase plus Dexmedetomidine plus Triamcinolone — transforaminal fluroscopic epidural injection
  Arms: dex plus hyalase group

SUMMARY:
use of dexmedtemodine to augment analgesia in cases of failed back surgery

ELIGIBILITY:
Inclusion Criteria:

* Age group. 25-75ys old
* Both sex.
* persistent (at least 6 month) pain and or disability following laminectomy with or without sensory-motor neurological deficits or any form of urinary or bowel incontinence
* Patients suffering from persistent (> 6 months) back pain following laminectomy for spinal canal stenosis and/or discectomy for herniated nucleus pulposus documented by magnetic resonance imaging (MRI) were included for screening and enrollment.

Exclusion Criteria:

* Diabetic patients.
* Refusal to participate
* MRI with disc sequestration, concurrent sacro-ilitis, facet arthropathy .
* Coagulopathic patients

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
pain assesment | 6 months
  visual analogue scale

SECONDARY OUTCOMES:
functional diability | 6 months
  Modified Oswestry Disability Questionnaire....0% to 20%: minimal disability:....21%-40%: moderate disability: 41%-60%: severe disability...61%-80%: crippled
acute complications | 6 hours after injection
  number of patients developed epidural hematoma by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, ALMinya, Minya Governorate, Egypt